CLINICAL TRIAL: NCT02004639
Title: Taiwan: Institutional Review Board
Brief Title: Trismus Prevention, Diagnosis and Management: Radiotherapy Planning, Early Detection, and Physical Therapy Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FEMH No.101127-F
Record Dates: First submitted 2013-11-28; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: IMRT or HT with chemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Mastictors sparing group (Active Comparator): Using IMRT or HT to do masticators sparing techniques and physical therapy to prevent trismus.
  Interventions: Radiation: Masticators sparing techniques
- Masticators not sparing group (No Intervention): The patients do not receive masticators sparing technique as traditional techniques but still receive physical therapy after radiotherapy to prevent trismus.
- EA group (Active Comparator): Using masticators sparing techniques and electro-acupunture stimulation to prevent trismus
  Interventions: Other: electro-acupunture treatment
- Sham-EA group (Sham Comparator): Using masticators sparing techniques but with sham EA stimulation.
  Interventions: Other: electro-acupunture treatment

INTERVENTIONS:
Radiation: Masticators sparing techniques
  Arms: Mastictors sparing group
Other: electro-acupunture treatment — electro-acupunture treatment and sham-EA
  Arms: EA group; Sham-EA group

SUMMARY:
Trismus Prevention, Diagnosis and Management: Radiotherapy Planning, Early detection, and Physical Therapy Intervention

DETAILED DESCRIPTION:
The optimal management of head and neck squamous cell carcinoma typically involves primary surgical resection, and the indications for adjuvant radiotherapy are based on pathologic markers of intermittent - and high-risk disease, which include positive margins, extracapsular nodal extension, lymphovascular invasion, and perineural invasion (1-3). Trismus is one of long term sequelae of radiotherapy for head and neck cancer patient. The prevalence of trismus after head and neck oncology treatment could be as high as 42% (4). It is significantly reducing nutrition due to impaired mastication (5). The loss of function appears to be related to damage and fibrosis to the muscles of mastication. Radiation therapy involving the temporomandibular joint, the pterygoid muscles, the temporalis or the masseter muscle is most likely to result in trismus (5, 6). Moreover, there may be scar tissue from radiation or surgery, nerve damage, or a combination of these factors (6, 7). In addition, the doses of RT levels in excess of 60 Gy (8) or the configuration of the radiation field increasing (9) are more likely to cause trismus. These data were documenting the clinical results of conventional radiotherapy (RT).

Recently, extensive data suggest that intensity-modulated radiation therapy (IMRT) is safe and efficacious in the adjuvant setting for oral cavity cancer (OCC) (10-12). Hsiung et al. (13) and Chen et al. (14) confirmed that radiation induced trismus progressed over time and improved by IMRT. Hsiung et al. (13) found the averages of normalized maximal interincisal distance (MID) were 94% and 98.1% at 5 ms and 12 ms post-IMRT, respectively. In addition, only 0.2 mm the deterioration of radiation-induced trismus in the period from 12-18 months post-IMRT was noted. Moreover, Chen et al. (14) also confirmed that radiation induced trismus progressed over time and improved by IMRT. However, Kent et al. (15) examined the incidence of trismus in IMRT group compared to conventional radiotherapy group. There was no significant difference in the maximum vertical dimension between the IMRT and the conventional RT groups, (38.8 ± 9.0 vs 33.7 ± 10.1 mm, respectively, p = 0.11).

Helical tomotherapy (HT) is conceptually regarded an image-guided IMRT. HT was designed and developed with advantages in sharper dose gradients and better normal tissue sparing. Our and the other clinical experience of using HT for locally advanced head and neck cancer had achieved encouraging results along with less toxicity, such lower percentage of dermatitis and xerostomia when compared with previous reports (16-18). HT provides better normal tissue sparing and sharper dose gradients than IMRT (19, 20).Chen et al. (19) compared HT and IMRT for nasopharyngeal carcinoma and noted that HT significantly reduced dose to the contralateral parotid gland and improved dose homogeneity to the PTVs. Additionally, HT reduced mean doses to brainstem (p = 0.02), larynx (p = 0.03), and oral cavity (p = 0.03). Similarly, for head-and-neck cancer, HT plans also provided favorably results compared with the step-and-shoot IMRT plans. They are expected to be able to reduce the parotid normal tissue (average 6.5 Gy) complication probability further, keeping similar target dose homogeneity (21). Furthermore, HT provided better mandible sparing than IMRT with mean dose decreased from 34.9 Gy (IMRT) to 30.7 Gy (HT) (20). However, can HT provide better normal tissue sparing to reduce the incidence of trismus? It's still an interesting issue to discuss.

In our 4-year initial clinical experience of 39 postoperative OCC patients treated with HT, we noted the incidences of grade 1 and grade 2, 3 trismus [according to the Common Terminology Criteria for Adverse Events v3.0 (CTCAE v3.0) ] appear inversely trend in time sequence with post-HT treatment (Fig. 1). These observations hint the possible of decreasing late complications of HT by better normal tissue sparing and sharper dose gradients (16-18) and responses to radiation induced trismus improved by IMRT (13, 14).

According to previous study (6), Magnetic resonance imaging (MRI) could provide advantage findings in masticator structures in patients with trismus developing after radiotherapy for nasopharyngeal carcinoma (NPC). The abnormalities comprising radiotherapy-induced masticator muscle fibrosis or inflammation, denervation atrophy of the masticator muscles secondary to mandibular nerve damage, osteoradionecrosis change of mandibular rami, perimasticator fibrosis extending into the masticator space and post RT damage of the parotid gland. The presence of several MRI abnormalities in the masticator structures of patients with trismus after radiotherapy suggests that trismus is multifactorial. However, there was no good correlation data between the severities of trismus with these image findings and thus these changes may possible due to non-specific inflammatory and fibrosis reactions after radiation. Also, there was no correlation data between radiation dosages with these abnormality, so all these findings may also result from other causes such as surgery or chemotherapy. Therefore, we try to evaluate MRI examinations performed in patients before and after trismus establishing following radiotherapy for OCC patients, in order to identify the range and frequency of underlying diseases that may cause this complication. We retrospect the OCC patients using MRI signal abnormality scores (SA score), separating the patient according to their clinical trismus grading into three groups, the mean SA score of grade 0 patient is 8.5, grade 1 is 6.76 and grade 2 is 4.87. Compared with group 2 patients, there are statistically significant differences between group 1 (p= .04) as well as group 0 (p= .02), respectively. It means the SA score could correspond to the trismus grade (Fig. 2).

Rehabilitation training can improve swallow function and slow down the progress of trismus in NPC patients following radiotherapy. The efficacy rate (percentage of patients with excellent or effective results) of rehabilitation group was higher than that of control group (77% vs. 43%), and the difference was statistically significant (p = 0.02). The efficacy rate of trismus in the rehabilitation group was significantly higher than that of the control group (64% vs. 28%, p = 0.02) (22). Using Therabite Jaw Motion Rehabilitation System (Therabite Corporation, Bryn Mawr, PA) for maintaining and/or improving mandibular range of motion in post-irradiated patients had been reported (23). They noted net increase in maximal interincisal distance ( MID) of Therabite group (13.6 mm [+/- 1.6 mm]) was significantly greater than unassisted exercise group (6.0 mm [+/- 1.8 mm]) and mechanically assisted mandibular mobilization with stacked tongue depressors combined with unassisted exercise group (4.4 mm [+/- 2.1 mm]) (P < .05) at week 6 and thereafter. These data supported the benefits of rehabilitation for trismus following RT. However, rehabilitation following new RT techniques have synchronic effect to improve patient's quality of life are another interesting points need to discuss.

Acupuncture is an ancient Chinese method to treat diseases and relieve pain. Electro-acupuncture (EA) is one of many physical measures used to relieve musculoskeletal pain and to improve the associated restricted range of motion. Furthermore, electrical stimulation via skin patch electrodes is as effective as EA. Low frequency (2 Hz) and high frequency (100 Hz) of EA selectively induces the release of enkephalins and dynorphins in both experimental animals and humans. Clinical studies suggest its effectiveness for the treatment of various types of pain and spinally induced muscle spasm (24). In addition, acupuncture-like stimulation exerts physiologic effects on the central nervous system, mediated presumably by muscle afferent fibers. The effects may be relevant to relief of muscle spasm and musculoskeletal pain, and restoration of mobility (25). Moreover, the combined method of acupuncture with pressure on otopoints (the combination group) was used to treat with facial spasm. The total effective rates of the combination group, the acupuncture group and the pressure on otopoints group were 95.4%, 92.1% and 62.5% respectively; and the cure rates were 38.4%, 15.8% and 5% respectively. The differences in results of the three groups indicated that the therapeutic effectiveness of the combined method of acupuncture with pressure on otopoints is better than the other two therapeutic methods (26).These data hit the potential benefits of combination of EA and physical therapy. Moreover, electrical stimulation via skin patch electrodes is as effective as EA (24). Therefore, the effects of physical therapy combined with skin patch electrodes with different frequency maybe better than physical therapy alone following CCRT or RT are another interesting issue to discuss. Therefore, we designed the current prospective measurement study with 3 years of follow-up to evaluate the incidence and severity of radiation-induced trismus after IMRT and HT following physical therapy with or without electrical stimulation via skin patch electrodes using MRI to assess relevant pretreatment factors, treatment-related factors, and dosimetric parameters.

Specific Aims:

For Year 1:

1. To clarify the optimal doses of each muscle for those who with mild or non-trismus treated by IMRT or HT with retrospective clinical data
2. To testify whether MRI findings can have good correlation with the radiation dose and also clinical severity of trismus.
3. To testify whether IMRT or HT plan can achieve the optimal doses by re-plan same patients with new constrains. .

For Year 2:

1. To clarify whether newly planning techniques of IMRT or HT can decrease the incidence and progression of trismus for head and neck patients.
2. To testify whether MRI findings can serve as predictors for trismus during follow.
3. To clarify whether adding rehabilitation can provide synchronous benefits for trismus following newly RT planning techniques.

For Year 3:

1. To clarify whether HT can provide better clinical results for decreasing trismus for head and neck patients than IMRT.
2. To clarify whether MR image abnormalities of head and neck patient after IMRT will change after early introduction of rehabilitation.
3. To clarify whether electrical stimulation via skin on specific points combined with rehabilitation can provide synchronous benefits than rehabilitation alone for trismus following newly RT planning techniques.

ELIGIBILITY:
Inclusion Criteria:

Head and neck cancer underwent surgery followed by postoperative IMRT or HT with or without chemotherapy

Exclusion Criteria:

Patients treated for recurrent squamous cell carcinomas of the oral cavity (including neck recurrences) are excluded from this analysis. -distance metastasis, previous received radiotherapy or concurrent chemoradation therapy are excluded from this analysis. Patients treated for recurrent squamous cell carcinomas of the oral cavity (including neck recurrences) are excluded from this analysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Time to trismus Progression | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan